CLINICAL TRIAL: NCT00004986
Title: Open Label, Multi-Center Evaluation of Nitazoxanide for the Treatment of Cryptosporidiosis in Subjects With AIDS in the United States
Brief Title: Safety and Effectiveness of Nitazoxanide for the Treatment of Cryptosporidiosis in AIDS Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 253C; RM-NTZ-99-003
Record Dates: First submitted 2000-03-16; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Cryptosporidiosis; Drug Evaluation; Antiprotozoal Agents; Treatment Failure; nitazoxanide
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; AIDS-Related Opportunistic Infections | interventions — nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide

SUMMARY:
The purpose of this study is to see if it is safe and effective to treat cryptosporidiosis in AIDS patients with nitazoxanide.

DETAILED DESCRIPTION:
Patients take nitazoxanide daily for 8 weeks with a dose escalation after the first 4 weeks. Patients return to the hospital for examinations every 2 weeks during the 8-week treatment period and 6-week follow-up. Nitazoxanide therapy is discontinued in patients showing a complete clinical and parasitologic response (therapeutic cure) after 8 weeks of treatment and in patients showing a therapeutic cure at two consecutive visits (Weeks 2 and 4 or Weeks 4 and 6). These patients undergo a physical examination including stool analysis for Cryptosporidium parvum oocysts and routine laboratory tests at Weeks 2, 4, and 6 after completion of nitazoxanide therapy. Patients who do not show a complete clinical and parasitologic response (therapeutic failure) after 8 weeks of treatment are allowed to remain on nitazoxanide therapy through the Open Label Compassionate Use of Nitazoxanide in Treatment of Cryptosporidiosis in AIDS Patients (UMD-95-009) protocol.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a CD4 cell count of 50 cells/mm3 or less.
* Have evidence of cryptosporidium infection in their stool sample within 10 days of study entry.
* Have watery stools at least three times a day at least 5 days a week for 21 days prior to enrollment.
* Are able to take medications by mouth.
* Are at least 13 years old (consent of parent or guardian required if under 18).
* Agree to use an effective method of birth control (such as condoms) during the study.

Exclusion Criteria

Patients will not be eligible if they:

* Have certain diseases or infections of the intestines.
* Have ever taken nitazoxanide.
* Have taken certain experimental drugs within 14 days of enrollment.
* Will need to take certain other medications during the study such as paromomycin, azithromycin, and clarithromycin.
* Have started a new anti-HIV therapy within 4 weeks of study entry or plan on starting one during the study.
* Are pregnant or breast-feeding.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2000-02

CONTACTS AND LOCATIONS:
Locations (1):
- Julie Ryner, Tampa, Florida, United States